CLINICAL TRIAL: NCT05037526
Title: Diabetes in Pregnancy Project Und Mobile Health in Gestational Diabetes: An Open Label Randomized Controlled Monocentric Trial on the Utility of Real Time Continuous Glucose Monitoring in the Care of Gestational Diabetes Versus Standard Care
Brief Title: Utility of Real Time Continuous Glucose Monitoring in the Care of Gestational Diabetes Versus Standard Care in Pregnancy Outcomes
Acronym: DiP GlucoMo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCB_GDMV4.0
Record Dates: First submitted 2021-07-29; First posted 2021-09-08 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexcom G System (Active Comparator): The Dexcom G6 or current version intended use is for the management of diabetes. It is a small flexible device that records interstitial glucose levels every 5 min and is intended to replace fingerstick blood glucose testing for diabetes treatment decisions. Interpretation of the Dexcom G6 or current version System results should be based on the glucose trends and several sequential readings over time. The system consists of a sensor, transmitter, receiver and mobile app.
  Interventions: Device: Dexcom G System
- Standard care of gestational diabetes with self monitoring blood glucose (SMBG) (Active Comparator): SMBG (self-monitoring of blood glucose) is recommended for women with gestational diabetes that involves finger pricking up to six times daily.
  Interventions: Device: Self monitoring blood glucose

INTERVENTIONS:
Device: Dexcom G System — Continuous glucose monitoring system
  Arms: Dexcom G System
Device: Self monitoring blood glucose — Standard Care
  Arms: Standard care of gestational diabetes with self monitoring blood glucose (SMBG)

SUMMARY:
Once a pregnant mother is diagnosed with gestational diabetes mellitus (GDM), she will be treated with either diet, medication (i.e., insulin), or both. The most important factor in GDM management is glycemic control to reduce adverse outcomes. Blood glucose levels have become the "key player" for monitoring and directing treatment during pregnancy. Large trials have confirmed that treatment of GDM to optimize glycemic control can decrease the incidence of many of these associated adverse maternal and neonatal outcomes. Up to now, SMBG (self-monitoring of blood glucose) is recommended for women with gestational diabetes that involves finger pricking up to six times daily. However, SMBG provides an incomplete picture of the daily glucose profile due to long intervals between finger pricking, and inaccurate self-reported measurements, which heavily rely on patients' compliance.

DETAILED DESCRIPTION:
The incidence of obesity and diabetes is rising worldwide even in younger populations. With a rise in maternal obesity also gestational diabetes mellitus (GDM) becomes more prevalent with a prevalence of up to 18% of pregnancies. Up to now, SMBG (self-monitoring of blood glucose) is recommended for women with gestational diabetes that involves finger pricking up to six times daily. The main purpose of this study is to prove that real time continuous glucose monitoring (rt-CGM) can effectively reduce the risk for adverse pregnancy and neonatal outcome in GDM. It is further hypothesized that rt-CGM can optimize maternal glycaemic control, increase patients satisfaction and adherence to management strategies of GDM. This is a open label randomized controlled trial with two parallel groups.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* GDM diagnosis between 24 0/7- 28 0/7 weeks of pregnancy by a 75g oral glucose test (oGTT)
* Maternal age of 18 to 45 years,
* Singleton gestation
* Gestational age ≥ 24 0/7 weeks and <32 0/7 weeks at enrollment.

Exclusion Criteria:

* Known hypersensitivity or allergy to the sensor
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders of the participant
* Participation in another study with investigational drug or product within the 30 days preceding and during the present study
* Maternal age < 18 years,
* Multi-fetal gestations,
* Known fetal structural or chromosomal anomalies
* Chronic use of medications associated with hyperglycemia (steroids)
* Planned preterm delivery
* Overt diabetes mellitus type 1 or 2
* HbA1c by study entry > 6.5%
* History of bariatric surgery or other surgeries that induce malabsorption
* Fetal growth restriction by study entry

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 302 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Composite adverse pregnancy and neonatal outcome | 2 years
  The primary endpoint is composite adverse pregnancy and neonatal outcome; the proportion of large for gestation age (LGA) newborns (birth weight >90th centile); fetal macrosomia (estimated fetal weight over the 95th centile); incidence of polyhydramnios (maximal vertical pocket ≥ 8 cm); rate of neonatal hypoglycaemia; occurrence of stillbirth. Every each and one of these variables contributes to a better neonatal outcome and are associated. This composite endpoint includes factors influencing decisive the neonatal outcome.

SECONDARY OUTCOMES:
Initiated Therapy | 10-14 weeks
  Need for antiglycemic therapy in example Insulin yes/no
Glycemic Outcomes 1 | 10-14 weeks
  Glycemic variability including number and duration of hypoglycemic and hyperglycemic events, mean interstitial glucose in mmol/L and its standard deviation (SD) A hypoglycemic event was defined for two separate analyses as excursions of at least 15 min below the target range (<3.5 mmol/L), and a hyperglycemic event was defined for two separate analyses as excursions of at least 15 min above the target range (>7.8 mmol/L).
Glycemic Outcomes 2 | 10-14 weeks
  Time in glucose target in %
Glycemic Outcomes 3 | 10-14 weeks
  Duration and frequency postprandial hyperglycaemic excursions
Glycemic Outcomes 4 | 10-14 weeks
  Hemoglobin A1c (HbA1c) values (at inclusion, birth and postpartum) in %
Pregnancy complications | 10-14 weeks
  Pregnancy Complications such as
  * Placenta insufficiency (Estimated fetal weight < 10th centile and blood flow changes),
  * Gestational hypertension (systolic blood pressure ≥ 140 mm Hg or diastolic blood pressure ≥ 90 mg Hg on two occasions at least 4 hours apart)
  * Preeclampsia (international Society for the Study of Hypertension in Pregnancy (ISSHP) definition)
Mode of Delivery | 10-14 weeks
  Mode of delivery including cesarean delivery, induction of labor, need for operative vaginal delivery (forceps or vacuum-assisted vaginal delivery)
Need for induction of labor | 10-14 weeks
  Induction of labor yes/no
Obstetrical outcome | 10-14 weeks
  Obstetric injury yes/no
Maternal outcomes | 10-14 weeks
  Body mass index (BMI) (pre-pregnancy and at the time of delivery) weight and height will be combined to report BMI in kg/m^2
Maternal weight gain | 10-14 weeks
  Weight gain after GDM diagnosis in kg
Maternal Compliance | 10-14 weeks
  Adherence to therapy yes/no
Maternal satisfaction questionnaire | 10-14 weeks
  Patient satisfaction after pregnancy evaluated through a questionnaire
Postpartum disorder | 10-14 weeks
  8 weeks postpartum oral glucose test values in mmol/L
Birth age | 10-14 weeks
  Gestational age at delivery in weeks
Preterm | 10-14 weeks
  Preterm delivery (delivery < 37 weeks gestational age) yes/no
Neonatal weight | 10-14 weeks
  Birth weight in grams
Neonatal outcome | 10-14 weeks
  Small for gestational age (birth weight < 10%) yes/no
Neonatal condition | 10-14 weeks
  Poor condition at birth (Apgar score at 5 minutes <7, Arterial pH of <7.0) yes/no
Neonatal Morbidity | 10-14 weeks
  Perinatal morbidity prior to hospital discharge.
Neonatal birth trauma | 10-14 weeks
  Birth trauma (brachial plexus injury, or clavicular, humeral, or skull fracture)
Resuscitation | 10-14 weeks
  Need for resuscitation yes/no
Neonatal Care | 10-14 weeks
  Admission to neonatal intensive care unit (NICU) with length of stay in days
Respiratory distress syndrome | 10-14 weeks
  Respiratory distress syndrome (need for supplemental oxygen > 4 hours after birth) yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Amylidi-Mohr, MD, Principal Investigator — Uniuversity Hospital and University of Bern
Locations (1):
- University Hospital of Bern, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Castorino K, Polsky S, O'Malley G, Levister C, Nelson K, Farfan C, Brackett S, Puhr S, Levy CJ. Performance of the Dexcom G6 Continuous Glucose Monitoring System in Pregnant Women with Diabetes. Diabetes Technol Ther. 2020 Dec;22(12):943-947. doi: 10.1089/dia.2020.0085. PMID 32324061
- [Result] Cosson E, Baz B, Gary F, Pharisien I, Nguyen MT, Sandre-Banon D, Jaber Y, Cussac-Pillegand C, Banu I, Carbillon L, Valensi P. Poor Reliability and Poor Adherence to Self-Monitoring of Blood Glucose Are Common in Women With Gestational Diabetes Mellitus and May Be Associated With Poor Pregnancy Outcomes. Diabetes Care. 2017 Sep;40(9):1181-1186. doi: 10.2337/dc17-0369. Epub 2017 Jul 19. PMID 28724718
- [Result] Feig DS, Donovan LE, Corcoy R, Murphy KE, Amiel SA, Hunt KF, Asztalos E, Barrett JFR, Sanchez JJ, de Leiva A, Hod M, Jovanovic L, Keely E, McManus R, Hutton EK, Meek CL, Stewart ZA, Wysocki T, O'Brien R, Ruedy K, Kollman C, Tomlinson G, Murphy HR; CONCEPTT Collaborative Group. Continuous glucose monitoring in pregnant women with type 1 diabetes (CONCEPTT): a multicentre international randomised controlled trial. Lancet. 2017 Nov 25;390(10110):2347-2359. doi: 10.1016/S0140-6736(17)32400-5. Epub 2017 Sep 15. PMID 28923465
- [Result] Inayama Y, Yamanoi K, Shitanaka S, Ogura J, Ohara T, Sakai M, Suzuki H, Kishimoto I, Tsunenari T, Suginami K. A novel classification of glucose profile in pregnancy based on continuous glucose monitoring data. J Obstet Gynaecol Res. 2021 Apr;47(4):1281-1291. doi: 10.1111/jog.14677. Epub 2021 Jan 27. PMID 33501738
- [Result] Polsky S, Garcetti R, Pyle L, Joshee P, Demmitt JK, Snell-Bergeon JK. Continuous glucose monitor use with and without remote monitoring in pregnant women with type 1 diabetes: A pilot study. PLoS One. 2020 Apr 16;15(4):e0230476. doi: 10.1371/journal.pone.0230476. eCollection 2020. PMID 32298269
- [Result] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Derived] Amylidi-Mohr S, Zennaro G, Schneider S, Raio L, Mosimann B, Surbek D. Continuous glucose monitoring in the management of gestational diabetes in Switzerland (DipGluMo): an open-label, single-centre, randomised, controlled trial. Lancet Diabetes Endocrinol. 2025 Jul;13(7):591-599. doi: 10.1016/S2213-8587(25)00063-4. Epub 2025 May 26. PMID 40441173